CLINICAL TRIAL: NCT04278495
Title: The Effect of Losartan on the Recoverability of Renal Function in Anuric and Oliguric Patients With Unilateral Obstructed Kidney: A Double Blind Randomized Placebo-controlled Trial
Brief Title: The Effect of Losartan on the Recoverability of Renal Function in Anuric and Oliguric Patients With Unilateral Obstructed Kidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOSARTAN.OBST.UROPATHY
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Losartan Adverse Reaction; Uropathy; Uropathy Obstructive
MeSH Terms: conditions — Urologic Diseases | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Active Comparator): to receive the medication Cozaar (Losartan Potassium 25mg "Merck Sharp & Dohme-UK"),
  Interventions: Drug: Cozaar (Losartan Potassium 25mg)
- Placebo (Placebo Comparator): to receive either placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cozaar (Losartan Potassium 25mg) — Cozaar (Losartan Potassium 25mg)
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Previous experimental studies concluded that angiotensin receptor blockers can ameliorate the harmful inflammatory and histological changes after relief of obstruction. Nevertheless, these witnessed effects have not been yet translated into the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* anuric and oliguric patients
* calculuar ureteral obstruction

Exclusion Criteria:

* anomalous kidney
* bilateral obstructed kidney
* history of recent use of angiotensin receptor blockers or angiotensin-converting enzyme inhibitors
* ASA score of >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Renographic glomerular filtration rate of the affected kidney. | 3 months
  assessed by radioisotope renography using 99mTc-mercaptoacetyltriglycine (99mTc-MAG3) in ml/min

SECONDARY OUTCOMES:
Serum creatinine change | 3 months
  assessed by serum creatnine in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shokier, Study Chair — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No